CLINICAL TRIAL: NCT06132711
Title: Safety and Efficacy of APRIL-BAFF-Bicephali CAR-T in Relapsed, Refractory Multiple Myeloma-A Single-center, Open-label, Single-arm Clinical Study
Brief Title: Safety and Efficacy of APRIL-BAFF-Bicephali CAR-T in Relapsed, Refractory Multiple Myeloma
Acronym: CAR-T
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xuzhou Medical University (Other)
Collaborators: Yake Biotechnology Ltd. (Industry)
Responsible Party: Principal Investigator, Kai Lin Xu，MD, professor, Xuzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XYFY2023-KL144-01
Record Dates: First submitted 2023-07-11; First posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Multiple Myeloma
Keywords: myeloma, Chimeric antigen receptor, April, TACI
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients treated with CAR T cells (Experimental): Peripheral blood mononuclear cells were collected and subjected to CD3+T cells were enriched, transfected with APRIL-BAFF-Bicephali lentiviral vector, expanded by in vitro culture, and pretreated with clear lymphocytes using the FC protocol before infusion of APRIL-BAFF-Bicephali CAR-T cells.
  Interventions: Other: APRIL-BAFF-Bicephali CAR-T cells

INTERVENTIONS:
Other: APRIL-BAFF-Bicephali CAR-T cells — Peripheral blood mononuclear cells were collected and subjected to CD3+T cells were enriched, transfected with APRIL-BAFF-Bicephali lentiviral vector, expanded by in vitro culture, and pretreated with clear lymphocytes using the FC protocol before infusion of APRIL-BAFF-Bicephali CAR-T cells.

SUMMARY:
This is a Single-center, open, single-arm clinical study, the goal of which was to evaluate the safety and efficacy of APRIL-BAFF-Bicephali CAR-T in relapsed and refractory multiple myeloma.The study consisted of four processes: patient enrollment screening; pre-CAR T cell therapy (including leukocyte apheresis, CAR T cell preparation and chemotherapy); inpatient monitoring phase for CAR T cell transfusion; and long-term follow-up phase

DETAILED DESCRIPTION:
This trial is a single-center, open, single-arm trial with a non-blinded design.

The study consisted of four processes: patient enrollment screening; pre-CAR T cell therapy (including leukocyte apheresis, CAR T cell preparation and chemotherapy); inpatient monitoring phase for CAR T cell transfusion; and long-term follow-up phase. The specific execution process is as follows:

1. Pre-enrollment assessment;
2. Patient enrollment and basic data collection;
3. Leukocyte apheresis and CAR-T cell production 3.1 Patients receive apheresis of about 12-15 liters to provide peripheral blood mononuclear cells for the preparation of CAR-T. In addition to the use of appropriate amounts of lymphocytes for CAR-T preparation, excess cells should be cryopreserved for subsequent studies and regulatory inquiries.

   3.2 APRIL-BAFF Bicephali CAR-T cell preparation. 4 cells were pretreated before transfusion Pretreatment was started-5 days before CAR-T cell revertant, and CAR-T cell treatment was performed 2 days after completion of chemotherapy. The purpose of chemotherapy is to reduce the tumor load on the one hand and to reduce the number of endogenous lymphocytes to facilitate the proliferation of reinfused CAR T cells. All patients were pretreated with FC regimen, fludarabine 30mg / m2 3days, cyclophosphamide 750mg / m2 1days. Antiemetic and symptomatic treatment could be given during chemotherapy, and generally treated with other chemotherapy.
4. Post-treatment assessment Subjects were assessed for toxicity as planned (weekly for 1 month, monthly for 6 months, and every 3 months thereafter); efficacy for every 4 weeks and every 3 months after 6 months. CAR-T cells were tested for in vivo expansion evaluation, including CD3 +, CD4 +, CD8 + T lymphocytes and B lymphocytes in peripheral blood.
5. purpose of research

1. Primary objective: To evaluate the effectiveness of APRIL-BAFF-Bicephali CAR-T in the treatment of relapsed and refractory multiple myeloma 2. Secondary objective: To evaluate its safety 3. Study design type, principles, and test procedures

ELIGIBILITY:
Inclusion Criteria:

The set subject inclusion criteria include multiple documents of multiple myeloma, no effective treatment options (e. g. autologous or allogeneic stem cell transplantation) and limited outcome (<2 years) with existing therapies, as follows:

1. Age is 18~70 years old;
2. Expected survival period of>12 weeks;
3. Multiple myeloma was diagnosed by physical examination, pathological examination, laboratory examination and imaging;
4. Patients with refractory multiple myeloma;
5. Patients with multiple myeloma recurrence;
6. ALT and AST <3 times normal; bilirubin <2.0mg / dl;
7. Quality of survival score (KPS)> 50%;
8. The patient has no serious heart, liver, kidney and other diseases;
9. Recurrence or no disease remission after hematopoietic stem cell transplantation or cellular immunotherapy;
10. Is not suitable for stem cell transplantation conditions or to abandon transplantation due to conditional restrictions;
11. Blood can be obtained intravenously, without other contraindications to leukapheresis;
12. Understand and voluntarily sign a written informed consent form.

Exclusion Criteria:

Exclusion criteria

1. Women who are pregnant or breastfeeding, or who have a pregnancy plan within six months;
2. Infectious diseases (such as HIV, active tuberculosis, etc.);
3. Active hepatitis B or hepatitis C infection;
4. Feasibility assessment screening demonstrated <10% transfection of targeted lymphocytes or underamplification under CD3 / CD28 co-stimulation (<5-fold);
5. Abnormal vital signs, and unable to cooperate with the examination;
6. Have mental or mental illness who cannot cooperate with the treatment and efficacy evaluation;
7. Highly allergic constitution or have a history of severe allergies, especially allergic to IL-2;
8. Subjects with a systemic infection or a severe local infection requiring anti-infective treatment;
9. Subjects with severe autoimmune disease;
10. The doctor believes there were other reasons for inclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events | :Baseline up to 28 days after CAR-T cells infusion]
  Adverse events assessed according to NCI-CTCAE v5.0

SECONDARY OUTCOMES:
overall response rate (ORR) | Month 6, 12, 18 and 24
  Assessment of ORR at Month 6, 12, 18 and 24
complete response (CR) | Month 6, 12, 18 and 24
  Assessment of CR at Month 6, 12, 18 and 24
Overall survival (OS) | Month 6, 12, 18 and 24
  Assessment of OS at Month 6, 12, 18 and 24
Event-free survival (EFS) | Month 6, 12, 18 and 24
  Assessment of EFS at Month 6, 12, 18 and 24

CONTACTS AND LOCATIONS:
Overall Officials: Kailin Xu MD, PD, Study Chair — The Affiliated Hospital oh Xuzhou Medical University
Locations (1):
- Kailin Xu, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No